CLINICAL TRIAL: NCT03019042
Title: Efficacy and Safety of Hou Gu Mi Xi in Patients With Spleen Qi Deficiency and Non-organic Gastrointestinal Disorders: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Hou Gu Mi Xi in Patients With Spleen Qi Deficiency and Non-organic Gastrointestinal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Collaborators: Nanchang Hongdu Hospital of Traditional Chinese Medicine (Unknown); Nanchang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhou, Lecturer, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JXUTCM-EBM-01
Record Dates: First submitted 2017-01-07; First posted 2017-01-12 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Gastrointestinal Disease
Keywords: Hou Gu Mi Xi; Shen Ling Bai Zhu San; mild gastrointestinal disorders; traditional Chinese medicine; randomized controlled trial
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hou Gu Mi Xi (Experimental): Patients in this arm receive Hou Gu Mi Xi, with oral dose of 30 g/day (contain 10.1 herb materials) during entire follow up period (2 years). HGMX is composed of 10 dietary Chinese herbs (including ginseng (Renshen), tuckahoe (Fuling), coixenolide (Yiyiren), Chinese yam (Shanyao), lotus seed (Lianzi), amomum (Sharen), platycodon (Jiegen), white hyacinth bean (Baibiandou), licorice (Gancao), and orange peel (Jupi)), early rice, and oats.
  Interventions: Dietary Supplement: Hou Gu Mi Xi
- placebo (Placebo Comparator): Patients in this arm receive placebo, with oral dose of 30 g/day during entire follow up period (2 years). The placebo is only consist of early rice and oats.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Hou Gu Mi Xi — Hou Gu Mi Xi is a dietary therapy form of Shen Ling Bai Zhu San, of which removes atractylodes and platycodon grandiflorum, adds perilla leaf for adapting a dietary therapy.
  Arms: Hou Gu Mi Xi
Other: placebo — The placebo has same appearance, taste and smell as Hou Gu Mi Xi.
  Arms: placebo

SUMMARY:
This trial aims to determine whether Hou Gu Mi Xi is an effective treatment for improving symptoms and indicators in patients with spleen qi deficiency and mild gastrointestinal disorder.

DETAILED DESCRIPTION:
Chronic gastrointestinal disorders are one of major health problems around the globe. The annual number of patients with chronic gastrointestinal disorders was about 60 to 70 million in American. According to the American statistics in 2014, 4.6 million admissions and 230 thousand patients died due to chronic gastrointestinal disorders. The direct or indirect costs caused by chronic gastrointestinal disorders reached at 142 billion dollars. In China, the incidence of chronic gastrointestinal disorders is 7.3‰ among urban residents, which ranks No. 5 among all diseases and leads to 975 dollars of annually medical costs for per patient.

Along with the development of medical science, traditional Chinese medicine (TCM) is playing an increasingly rule in treatment of chronic gastrointestinal disorders, especially for these mild gastrointestinal disorders which are hard to obtain efficacy in western medicine. Shen Ling Bai Zhu San, a classic Chinese medicinal formulae originally described in Tai Ping Hui Min He Ji Ju Fang in the Fang Song Dynasty (1102 AD), is composed of ginseng, tuckahoe, atractylodes, baked licorice, coixenolide, Chinese yam, lotus seed, shrinkage fructus amomi, platycodon grandiflorum, white hyacinth bean, and dried orange peel. It has effects of replenishing qi and invigorating spleen (spleen is a TCM conception different from western medicine), as well as penetrating wet and antidiarrheal. It is mainly used for treating the syndrome of spleen qi deficiency, including dyspepsia, chest and stomach distress, borborygmus and diarrhea, limb weakness, thin body, sallow complexion, pale tongue with white and greasy coating, and weak and slow pulse, etc. In the theory of TCM, spleen is the source for producing qi and blood and thus is the root of life. Shen Ling Bai Zhu San could invigorate spleen by supplying spleen and remove wet, and finally nourish the stomach and intestine.

To date, Shen Ling Bai Zhu San is mainly used to treat mild gastrointestinal disorder like irritable bowel syndrome and functional dyspepsia in patients with a TCM syndrome of spleen qi deficiency. Pharmacologic study revealed that Shen Ling Bai Zhu San could adjust function of anaerobic and aerobic bacteria in gastrointestinal tract; specifically, it could improve the proliferation of probiotics (such as bifidobacterium) and inhibit the main resistance strains (such as enterococcus) and thus has an effect to improve gastrointestinal symptoms.

Hou Gu Mi Xi is a dietary therapy form of Shen Ling Bai Zhu San, of which removes atractylodes and platycodon grandiflorum (two herbs that could not be used as food) from Shen Ling Bai Zhu San, and adds perilla leaf for adapting a dietary therapy. Hou Gu Mi Xi used the main formula of Shen Ling Bai Zhu San, so that it could theoretically maintain the treatment effects. Although the reliable health effects of Shen Ling Bai Zhu San has been proved in previous studies, Hou Gu Mi Xi is optimized in formula and its preparations changed from electuary to rice paste, so that its functional mechanism and efficacy may also be different. Therefore, the investigators plan to perform a hospital-based randomized controlled trial, enroll patients from five hospitals in Nanchang City of Jiangxi Province in China, for assessing efficacy and safety of Hou Gu Mi Xi on Gastrointestinal symptoms and indicators in Patients with Spleen Qi Deficiency and Mild Gastrointestinal Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patient should have mild gastrointestinal disorder without any organic pathologic changes (see exclusion criteria) by diagnosis of gastroscopy within 6 months, which mainly include chronic non-atrophic gastritis, functional gastrointestinal disorders, irritable bowel syndrome, and functional dyspepsia
* Patient should be status of spleen qi deficiency, that is, meet 2 main symptoms of spleen deficiency and 2 main symptoms of qi deficiency, or have 2 main symptoms of spleen deficiency, 1 main symptoms of qi deficiency and 1 tongue symptom, or have 1 main symptom of spleen deficiency + 1 main symptom of qi deficiency + 2 secondary symptom + 1 tongue symptom as follow:

  1. Main symptoms of spleen deficiency: a) poor appetite; b) abnormal stool (loose, diarrhea); c) abdominal distention after meal or afternoon
  2. Main symptoms of qi deficiency: a) fatigue; b) tired mind and taciturnity
  3. Secondary symptoms: a) tastelessness, hypodipsia, like hot drink, or polysialia; b) abdominal pain, as a result either patients like warm or press, or remit after meal, or occur when work; c) nausea and vomiting; d) fullness in stomach; e) abnormal bowel sounds; f) lean or puffiness; g) sallow complexion; h) powerless defecation weakness; i) edema
  4. Tongue symptoms: pale or swollen or teeth-printed tongue with thin and white fur
* Fourteen years old or more
* Sign the informed consent

Exclusion Criteria:

* Patients who have organic pathologic changes, including peptic ulcer, gastrointestinal erosions, gastroesophageal reflux disease, acute gastrointestinal hemorrhage or perforation, structural changes in gastrointestinal structure, gastrointestinal vascular diseases, ileus, and benign tumor
* Pregnancy or breast-feeding women
* Allergic to sample or sample composition
* impaired liver function, including one of following condition: a) total bilirubin > 2 upper limit of normal (ULN); b) alanine transaminase >2 ULN; or c) aspartate aminotransferase >2 ULN
* impaired kidney function, that is, serum creatinine >2 ULN
* obviously abnormal electrocardiogram
* patients who undertaken drugs that could cause damage in stomach and intestine, or patients experience side effects of dyspepsia as undertaking non-steroidal anti-inflammatory drugs, theophylline, oral antibiotic or potassium supplements within 3 months
* patients who are receiving any agents or other intervention for treating his/her gastrointestinal disorder
* patients with any malignant tumor
* patients who have severe mental disorders so that could not control his/her action and coordinate the treatment in this trial.
* patients who are unwilling to provider personal information and enter this trial
* patients who cannot understand and sign informed consent

Ages: 14 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total scores of Spleen Qi Deficiency Symptoms Grading and Quantifying Scale (Units on a scale) | At baseline and 2, 4, 8, 26, 52, 78 and 104 weeks
  Higher score indicates severer symptoms of Spleen Qi Deficiency. Units of measure (Units on a scale)

SECONDARY OUTCOMES:
Change from baseline in Gastrin-17 (ng/L) | At baseline and 52 and 104 weeks
  To determine whether the interventions improve gastric function
Quantitative results of gastroscopy | At baseline and 104 weeks
  To assess pathologic changes
Changes from baseline in body weight (kg) | At baseline and 52 and 104 weeks
  To determine whether the interventions improve body weight
Changes from baseline in body mass index (kg/m2) | At baseline and 52 and 104 weeks
  To determine whether the interventions improve body mass index
Incidence of any adverse events | From the first dose of intervention up to 104 weeks
  Assessing by abnormal results (indicated by more or less than 2 × normal reference interval) in the routine blood, urine, and stool tests, liver function tests (alanine transaminase [ALT], aspartate aminotransferase [AST], total bilirubin [TBIL], direct bilirubin [DBIL], indirect bilirubin [IBIL]), kidney function tests (serum creatinine [SCr] and urea nitrogen [BUN]), and electrocardiogram as well as doctor-evaluated and patient-reported adverse events
Incidence of severe adverse events | From the first dose of intervention up to 104 weeks
  AEs that lead to new or prolonged hospitalization, disability, admission to intensive care unit, life danger, and death
Incidence of drug-related adverse events | From the first dose of intervention up to 104 weeks
  This outcome is assessed by blinded clinicians in each research center
Incidence of withdrawn due to adverse events | From the first dose of intervention up to 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Zhu, Ph.D., Study Chair — Jiangxi University of Traditional Chinese Medicine
Locations (1):
- Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data are not planned to share.

REFERENCES:
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States part I: overall and upper gastrointestinal diseases. Gastroenterology. 2009 Feb;136(2):376-86. doi: 10.1053/j.gastro.2008.12.015. Epub 2009 Jan 3. No abstract available. PMID 19124023
- [Background] Farthing M, Roberts SE, Samuel DG, Williams JG, Thorne K, Morrison-Rees S, John A, Akbari A, Williams JC. Survey of digestive health across Europe: Final report. Part 1: The burden of gastrointestinal diseases and the organisation and delivery of gastroenterology services across Europe. United European Gastroenterol J. 2014 Dec;2(6):539-43. doi: 10.1177/2050640614554154. No abstract available. PMID 25452850
- [Background] Wu TH, Chen IC, Chen LC. Antacid effects of Chinese herbal prescriptions assessed by a modified artificial stomach model. World J Gastroenterol. 2010 Sep 21;16(35):4455-9. doi: 10.3748/wjg.v16.i35.4455. PMID 20845514
- [Background] Yin GY, Chen Y, Shen XJ, He XF, Zhang WN. Study on the pathophysiologic basis of classification of 'spleen' deficiency in chronic gastritis. Chin Med J (Engl). 2005 Mar 20;118(6):468-73. PMID 15788127
- [Background] Yin GY, Zhang WN, Shen XJ, He XF, Chen Y. Study on the pathological basis of classification of spleen deficiency in chronic gastritis. Chin Med J (Engl). 2004 Aug;117(8):1246-52. PMID 15361303
- [Derived] Chen X, Nie H, Liu W, Zhou X, Nie J, Xie B, Chen D, Jiang Y, Zhang K, Fu Y, Yang D, Xiong Y, Zhao Z, Sun X, Zhu W. Efficacy and Safety of Hou Gu Mi Xi on Spleen Qi Deficiency in Patients with Nonorganic Gastrointestinal Disorders: Protocol for a Multicenter, Randomized, Placebo-Controlled Trial. Evid Based Complement Alternat Med. 2018 Dec 2;2018:1980491. doi: 10.1155/2018/1980491. eCollection 2018. PMID 30622590